CLINICAL TRIAL: NCT05003115
Title: MoVE: Motivational Strategies To Empower African Americans To Improve Dialysis Adherence
Brief Title: Motivational Strategies To Empower African Americans To Improve Dialysis Adherence
Acronym: MoVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ebele Umeukeje, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 211127 - MoVE; 5R03DK129626-02 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Dialysis treatment adherence; Hemodialysis; African American
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care
- Intervention (Experimental): Motivational interviewing intervention
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — In this trial, motivational interviewing (MI) is the intervention. The MI sessions will embody the spirit of MI (PACE - Partnership, Acceptance, Compassion and Evocation) and the use of MI strategies (OARS - Open-ended questions, Affirmations, Reflections and Summaries) and MI communication processes (engagement, focusing, evoking and planning).
  Other Names: MI
  Arms: Intervention

SUMMARY:
This study addresses the need to rigorously advance the science and understanding of the development, feasibility, acceptability and adoption of novel culturally-sensitive motivational strategies to improve dialysis treatment adherence among African Americans with end-stage kidney disease (ESKD). This study specifically aims to:

1. Gain advanced skills in the development and implementation of novel culturally sensitive motivational strategies
2. Acquire critical preliminary data for an R01-funded phase II efficacy trial testing the use of these motivational strategies to improve dialysis treatment adherence.

DETAILED DESCRIPTION:
Hemodialysis treatment non-adherence is a public health issue because of its association with excessive hospitalizations, high morbidity, mortality, and increased financial costs. Compared to whites, African Americans have a four-fold higher prevalence of end stage kidney disease (EKSD), higher non-adherence rates to hemodialysis, and higher odds of hospitalizations. Motivational interviewing, an evidence-based intervention that creates a bond between patients and providers, targets improvement in motivation-related psychosocial factors associated with adherence behaviors. Interventions for such factors are typically developed based on the dominant culture and may not be valid and generalizable to minority groups. Culturally tailored interventions lead to more durable change in African Americans yet there is a lack of studies testing the efficacy of such approaches to improve hemodialysis treatment adherence in African Americans. Use of culturally tailored motivational interviewing in African Americans with ESKD will promote health equity by improving dialysis treatment adherence, reducing hospitalizations, and enhancing other critical outcomes.

Our long-term goal is to establish culturally sensitive strategies and multi-level interactions to improve outcomes in kidney disease. The overall objective of this project is to evaluate the efficacy of a culturally tailored motivational interviewing intervention developed using a rigorous theoretical framework on improving hemodialysis treatment adherence in African Americans with ESKD. The central hypothesis is that culturally tailored motivational interviewing will lead to improved hemodialysis treatment adherence. We will test this hypothesis in the following Specific Aims in a randomized clinical trial (RCT) in African American patients with ESKD. Compared to usual dialysis care, we aim to: Evaluate the efficacy of 8 weeks of culturally tailored motivational interviewing (MoVE) on improving hemodialysis adherence at (1) 3 months, and (2) 6 months post-randomization. At the successful completion of the proposed research, the expected outcomes will include evidence of the efficacy of culturally tailored motivational interviewing on improving hemodialysis treatment adherence in African American patients with ESKD. The proposed research is innovative because of the novel application of a culturally tailored, evidence-based behavioral intervention developed using a rigorous theoretical network (PEN-3); the use of specifically-trained health coaches to optimize the intervention delivery; and the focus on understanding and overrepresented African American patients with ESKD to address the public health issue of hemodialysis treatment of non-adherence. Study results will provide a strong basis for conducting an effectiveness and implementation trial, which is expected to have a significant impact on hemodialysis adherence, hospitalizations, morbidity, and mortality. This research strongly aligns with NIDDK's mission to promote health equity by addressing health disparities in kidney disease.

Hemodialysis treatment non-adherence is an important modifiable contributor to end stage kidney disease (ESKD), with critical public health relevance to patients, providers, and health systems due to its association with excessive hospitalizations, exorbitant financial burden, and increase morbidity and mortality. Compared to Whites, African Americans ESKD patients have a four-fold higher ESKD prevalence, persistently higher hospitalization and rehospitalization risk, and higher rates of dialysis treatment non-adherence. The goals of this proposal are to: (1) evaluate the efficacy of culturally tailored motivational interviewing on improving hemodialysis treatment adherence in African Americans; (2) provide a strong basis for conducting a future effectiveness and implementation trial using evidence-based, culturally tailored motivational interviewing intervention to improve hemodialysis adherence, and reduce hospitalizations, morbidity, mortality, and exorbitant financial burden associated with dialysis treatment non-adherence; and (3) promote health equity by reducing existing health disparities and optimizing outcomes in ESKD.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Receiving hemodialysis treatments
* Been on hemodialysis for more than 30 days
* 18 years of age and older
* Within a 3-month look back at the time of screening, patients who have missed at least one dialysis session or shortened at least one dialysis session by 15 minutes.

Exclusion Criteria:

* Not self-identified as African American
* Impaired with mental status or severe illness
* Non-English speaking
* No documented evidence of dialysis treatment non-adherence
* Missed or shortened treatments due to hospitalizations or excused travel
* Terminal condition
* Living in a nursing home/rehab
* Planned transplant within the next 3 months
* Planned conversion to peritoneal dialysis within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebele M Umeukeje, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Vanderbilt Dialysis Clinic, Nashville, Tennessee
  - Vanderbilt Dialysis Clinic East, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard Care
Period: Overall Study
Arm/Group | Control | Intervention
Started | 15 | 14 (This reflects the total number of participants whose data was included in the analysis for the intervention, even if they dropped out of the study and did not complete the MI sessions and/or the surveys.)
Completed | 15 | 11
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57 [44 to 64] | 57 [46 to 63] | 57 [45 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
Adherence [Median (Inter-Quartile Range); unit: percentage of minutes completed] — Percentage of prescribed minutes attended in dialysis sessions not canceled for travel or hospitalization
  percentage of minutes completed | 94.43 [87.01 to 96.29] | 94.64 [86.99 to 99.07] | 94.54 [86.77 to 96.87]
Perceived Kidney Disease Self-Management Scale [Median (Inter-Quartile Range); unit: units on a scale] — The Perceived Kidney Disease Self-Management Scale (PKDSMS), is a measure to assess how dialysis patients view their self-efficacy in regard to dialysis treatment adherence. Four of the items (#s 1, 2, 6, 7) are reversed-scored. The score is the sum of the 8 individual items. The total PKDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's (dialysis).
  units on a scale | 35 [32 to 40] | 30 [26 to 36] | 32 [26 to 38]
Perceived Expectancies Index [Median (Inter-Quartile Range); unit: units on a scale] — The Dispositional Optimism items are #s 1, 3, 5, & 7; The Perceived Competence items are #s 2, 4, 6, & 8. Items # 2, 5, 6, & 7 need to be reverse scored. The overall score is calculated by summating the scores after reverse scoring 2,5,6, and 7. The score ranges from 8-48 with 48 being the highest perceived expectancies. The score can also be broken down into the above scales.
  units on a scale | 39 [31 to 44] | 39 [33 to 42] | 39 [32 to 44]
Life Orientation Test - Revised [Median (Inter-Quartile Range); unit: units on a scale] — Change in optimism will be measured by the 10-item Life Orientation Test - Revised (LOT-R) questionnaire which assesses individual differences in generalized optimism versus pessimism. Only 6 of the 10 items on the revised LOT are used to derive an optimism score. Of the 6 survey questions utilized, each question ranges in score from 1 to 5. Thus, scores in principle can range from 6 to 30. The scale is a continuous dimension of variability between optimism and pessimism with higher scores indicating high optimism (low pessimism) and lower scores indicating high pessimism (low optimism).
  units on a scale | 24 [18 to 25] | 24 [19 to 26] | 24 [18 to 25]
Healthcare Climate Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Change in autonomy support will be measured by the 6-item Health Care Climate (HCC) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous support, and higher scores reflect greater autonomous support. Population: Only 14 control participants were captured for this survey.
  units on a scale
    number analyzed (Participants) | 14 | 14 | 28
    (all) | 7.0 [6.6 to 7.0] | 5.3 [4.4 to 6.1] | 6.3 [5.0 to 7.0]
Autonomous Regulation [Median (Inter-Quartile Range); unit: units on a scale] — Change in autonomous regulation will be measured by the 6-item Autonomous Regulation (AR) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous regulation, and higher scores reflect greater autonomous regulation
  units on a scale | 7.0 [6.8 to 7.0] | 6.8 [6.1 to 7.0] | 7.0 [6.7 to 7.0]
Apathy Evaluation Scale [Median (Inter-Quartile Range); unit: units on a scale] — Change in apathy will be measured by the 7-item Apathy Evaluation Scale survey (AES-S) which measures three domains of apathy: deficits in goal-directed behavior; a decrement in goal-related thought content; and emotional indifference with flat affect. Each question ranges in score from 1 to 4. Item 3 is reverse-scored and then the sum of the 7 item scores is calculated. Range of scores is 7-28, with higher scores indicating more apathy.
  units on a scale | 26 [22 to 28] | 25 [24 to 27] | 26 [22 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Dialysis Treatment Adherence
Description: Abstraction of dialysis treatment adherence data from the dialysis units' records which includes data on every treatment that occurred or should have occurred within the time frame. Records will reflect dialysis treatments which were completed, shortened, missed or did not occur due to hospitalizations, ER visits or travel.
Time Frame: Week 8, i.e. the maintenance phase, days 31 through 60 post-randomization
Measure: Median (Inter-Quartile Range); unit: percentage of minutes completed
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 14
percentage of minutes completed | 95.85 [85.19 to 99.37] | 93.26 [80.35 to 99.01]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.101, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -6.36, 95% CI 2-sided [-14.17 to 1.44]

2. Secondary Outcome: Change in Autonomous Regulation
Description: Change in autonomous regulation will be measured by the 6-item Autonomous Regulation (AR) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous regulation, and higher scores reflect greater autonomous regulation
Time Frame: Week 8
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 of those completed the AR survey - the remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 7.0 [7.0 to 7.0] | 6.8 [6.4 to 7.0]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.78, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -0.10, 95% CI 2-sided [-0.79 to 0.59]

3. Secondary Outcome: Change in Autonomy Support
Description: Change in autonomy support will be measured by the 6-item Health Care Climate (HCC) questionnaire. Questions range in score from 1 to 7, and overall score is a mean of all items (range 1 - 7). Lower scores reflect less autonomous support, and higher scores reflect greater autonomous support.
Time Frame: Week 8
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 participants completed the (HCC) questionnaire. The remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 7.0 [6.8 to 7.0] | 5.2 [4.4 to 6.0]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.314, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -0.95, 95% CI 2-sided [-2.83 to 0.94]

4. Secondary Outcome: Change in Perceived Competence
Description: Change in perceived competence will be measured by the 8-item Perceived Kidney Disease Self-Management Scale (PKDSMS) questionnaire.Each question ranges in score from 1 to 5. Four of the items (#s 1, 2, 6, 7) are reversed-scored. The score is the sum of the 8 individual items. The total PKDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's (dialysis).
Time Frame: Week 8
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 participants completed the (PKDSMS) questionnaire. The remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 38 [35 to 40] | 34 [32 to 36]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.679, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -1.04, 95% CI 2-sided [-6.00 to 3.92]

5. Secondary Outcome: Change in Apathy
Description: Change in apathy will be measured by the 7-item Apathy Evaluation Scale survey (AES-S) which measures three domains of apathy: deficits in goal-directed behavior; a decrement in goal-related thought content; and emotional indifference with flat affect. Each question ranges in score from 1 to 4. Item 3 is reverse-scored and then the sum of the 7 item scores is calculated. Range of scores is 7-28, with higher scores indicating more apathy.
Time Frame: Week 8
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 participants completed the (AES-S) survey. The remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 26 [24 to 28] | 26 [23 to 28]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.994, Regression, Linear; Mean Diff. Adjusting for Baseline Values = 0.01, 95% CI 2-sided [-2.23 to 2.25]

6. Secondary Outcome: Change in Optimism
Description: Change in optimism will be measured by the 10-item Life Orientation Test - Revised (LOT-R) questionnaire which assesses individual differences in generalized optimism versus pessimism. Only 6 of the 10 items on the revised LOT are used to derive an optimism score. Four of the items are filler items and are not used in scoring. Of the 6 survey questions utilized, each question ranges in score from 1 to 5. Thus, scores in principle can range from 6 to 30. There are no 'cut-offs' for optimism or pessimism; the scale is a continuous dimension of variability between the two with higher scores indicating high optimism (low pessimism) and lower scores indicating high pessimism (low optimism).
Time Frame: Week 8
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 participants completed the (LOT-R) questionnaire. The remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 24 [22 to 26] | 22 [21 to 24]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.258, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -1.22, 95% CI 2-sided [-3.33 to 0.89]

7. Secondary Outcome: Perceived Expectancies Index
Description: The Dispositional Optimism items are #s 1, 3, 5, & 7; The Perceived Competence items are #s 2, 4, 6, & 8. Items # 2, 5, 6, & 7 need to be reverse scored. The overall score is calculated by summating the scores after reverse scoring 2,5,6, and 7. The score ranges from 8-48 with 48 being the highest perceived expectancies. The score can also be broken down into the above scales.
Time Frame: 8 Weeks
Population: 14 participants were reflected in the intervention arm of the participant flow module. Only 12 participants completed the survey. The remaining 2 dropped out of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 12
score on a scale | 43 [37 to 45] | 40 [34 to 44]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.857, Regression, Linear; Mean Diff. Adjusting for Baseline Values = -0.40, 95% CI 2-sided [-4.75 to 3.96]

ADVERSE EVENTS:
Time Frame: 6 months
Description: If a patient experienced an adverse event during the study, then the health coach or research assistant would notify the PI immediately , who would follow-up with the patient directly.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT05003115/Prot_001.pdf
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT05003115/SAP_002.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT05003115/ICF_003.pdf